CLINICAL TRIAL: NCT06623071
Title: Accupower ® HBV Performance Evaluation Quant Kit Bioneer Existation™FA 96/384
Brief Title: Accupower ® HBV Performance Evaluation Quant Kit Bioneer Existation FA 96/384
Acronym: BIOPERF-HBV
Status: Recruiting | Type: Observational
Sponsor: CerbaXpert (Other)
Collaborators: Bioneer Corporation (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2024-A01285-43; 2024-A01285-43 (Other: ANSM)
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-09

CONDITIONS: Hepatitis B
Keywords: HBV
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Evaluation performance in vitro medical device study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Infected patients: Patients infected with hepatitis B virus

SUMMARY:
As part of the CE marking of a hepatitis B diagnostic kit, the South Korean manufacturer Bioneer wishes to set up a performance study in France in accordance with the IVDR (RE 2017/746).

Cerba Xpert CRO of the Cerba Healthcare group promoted this performance study by setting up a prospective collection of blood samples from patients with hepatitis B virus and whose viral load is positive. This prospective collection will be carried out in 3 laboratories of the Cerba Healthcare group.

DETAILED DESCRIPTION:
Viral hepatitis are primarily human systemic infections caused by viruses hepatic diseases which cause damage to the liver by hepatocyte infection of the virus and/or a host immune response to the virus. (1) Hepatitis is grouped into five types (A, B, C, D, E) and is mainly transmitted by parenteral, sexual and fetomaternal. (2) Hepatitis B virus (HBV) was discovered in 1965 in the United States.(3)It is a DNA virus that belongs to the family Hepadnaviridae. (4) Hepatitis B infection is characterized by signs clinical conditions such as jaundice, asthenia, anorexia but in the vast majority of cases (98% of infections). The course of hepatitis B is not serious; Nine out of ten people will clear the virus thanks to their immune defenses: they heal spontaneously and are immune because they made antibodies against HBV.(5) In 10% of infected people (15% in men, 5% in women), the hepatitis virus B will remain in the liver where it will be more or less active. This activity leads to chronic hepatitis.

Approximately 316 million people are chronic carriers of HBV worldwide (1-3) and approximately 887,000 deaths are linked to the hepatitis B virus each year. Appropriate support for carrying Chronic HBV reduces the risk of transmission. The WHO has set the goal of elimination of viral hepatitis B and C in 2030.(5) The biomarkers specifically associated with this infection are: Hbs antigen (HbsAg), antibodies anti-Hbs, anti-HBc antibodies, Hbe antigen, anti-HBe antibodies, virus DNA in plasma.

Chronic hepatitis B is defined by the maintenance of HBs antigen in the blood beyond 6 months.(6) The diagnosis of acute hepatitis B is based on the combination of a clinical picture such as acute febrile state.

accompanied or followed by jaundice or an increase in hepatic transaminases (AST, ALT, gammaGT) and the presence of HBs antigen and anti-HBc IgM and viral DNA in the blood.(6) Treatment monitoring of chronic hepatitis B is carried out by monitoring the viral load of hepatitis B in the blood. Furthermore, quantification of viral load during hepatitis monitoring Chronic B is essential in order to be able to assess and anticipate the risk of progression towards fibrosis.(6) On the European market, quantitative determination of hepatitis B viral load as part of Diagnosis and monitoring of the disease is done by real-time PCR which is the reference technique.(7) As part of routine care, there are several diagnostic PCR kits that can be used on plasma or serum. Today, there are no CE approved PCR kits that allow the quantification of viral DNA at the both serum and plasma. Our study will make it possible to evaluate the performance of the Bioneer kit PCR kit AccuPower® Quant Kit Bioneer ExiStation™FA 96/384 on serum and plasma from patients with hepatitis B.

ELIGIBILITY:
Inclusion Criteria:

The patient to be included in this study must be able to understand the purpose research, in order to give free and informed consent.

* Subject aged over 18
* Subject presenting himself at the investigation center and responding to one of these two criteria:

  * Subject presenting with a prescription for determination HBV viral load
  * Subject with previously confirmed HBV infection by CE marked tests.
* Subject capable of understanding the aim of the research having given express free and informed consent
* Subject affiliated to or beneficiary of a social security system

Exclusion Criteria:

Protected subject: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial decision or administrative

• Subject participating in another clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Infected patients with hepatitis B virus
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Commutability between serum and plasma hepatitis B viral load results with the ACCUPOWER HBV Quant Kit Bioneer Existation™FA 96/384 | 4 months
  The submitted protocol is carried out as part of a 'commutability' study, that is to say for Compare two matrix types on the Accupower ® HBV Quant Kit Bioneer Existence™FA 96/384. Indeed, for these two matrices to be claimed in the IFU of the kit it is necessary to prove that the two matrices give the same result.
  The planned size of the evaluable cohort is 45 patients included over a period of 4 month. This size is justified by the recommendations of the applicable CLSI EP09 guide.
  This guide details the use of several mathematical models that guarantee robust analysis even on a small cohort size. The operating methodology of the results is detailed below, taken from the recommendations of the CLSI EP09 guide

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Cerba Xpert, Frépillon, Ile de Franace
  - Cerballiance Chemin vert, France, Paris

IPD SHARING:
Plan to Share IPD: No